CLINICAL TRIAL: NCT00002874
Title: A PHASE III TRIAL OF RADIATION THERAPY WITH OR WITHOUT CASODEX IN PATIENTS WITH PSA ELEVATION FOLLOWING RADICAL PROSTATECTOMY FOR pT3N0 CARCINOMA OF THE PROSTATE
Brief Title: Radiation Therapy With or Without Bicalutamide for Recurrent pT3N0 Prostate Cancer After Radical Prostatectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RTOG-9601; CDR0000065158; RTOG-R9601
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bicalutamide (Experimental): Radiation therapy + bicalutamide
  Interventions: Drug: bicalutamide; Radiation: radiation therapy
- Placebo (Placebo Comparator): Radiation therapy + placebo
  Interventions: Radiation: radiation therapy; Drug: placebo

INTERVENTIONS:
Drug: bicalutamide — One (150 mg) tablet by mouth daily for two years beginning immediately upon, or just prior to, the initiation of irradiation.
  Other Names: Casodex
  Arms: Bicalutamide
Radiation: radiation therapy — 64.8 Gy in 36 fractions (1.8 Gy in 5 daily sessions per week) to the original prostate volume, the tumor resection bed, and the proximal membranous urethra.
Drug: placebo — One tablet by mouth daily for two years beginning immediately upon, or just prior to, the initiation of irradiation.
  Arms: Placebo

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Androgens can stimulate the growth of prostate cancer cells. Hormone therapy using bicalutamide may fight prostate cancer by reducing the production of androgens. It is not yet known if radiation therapy is more effective with or without bicalutamide for prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy with or without bicalutamide in treating patients who have stage II or stage III prostate cancer and elevated prostate-specific antigen (PSA) levels following radical prostatectomy.

ELIGIBILITY:
Conditions for Patient Eligibility:

* The patient on entry will have no clinical evidence of disease by physical exam or by imaging studies. A positive ProstaScint scan alone without a confirmatory biopsy must not be used to exclude a patient. Eligible patients will be those who have undergone a radical prostatectomy (either retropubic or perineal) and pelvic lymphadenectomy (either open or laparoscopic) for carcinoma of the prostate, pathologic stage T3N0, or pT2 pN0 with positive inked resection margin, at least 12 weeks prior to study entry.
* Pathological T2 patients without positive margins, who are also pathologic N0 with prostatic fossa/anastamosis biopsy at the time of rising PSA documenting recurrent cancer, are eligible.
* At entry, the PSA must be between 0.2 and 4.0ng/ml, inclusive.
* A post-prostatectomy radioisotopic bone scan which was done within 16 weeks prior to entry must reveal no evidence of metastatic disease.
* Patient must be evaluated by both the radiation oncologist and the urologist prior to entry and judged to be a suitable candidate for radiation and hormonal therapy.
* Patient must have Karnofsky performance status >= 80.
* Patients must have a life expectancy in excess of 10 years.
* Patients must have, within 6 weeks prior to entry, a hemoglobin (Hgb) of >=10 gm, a white blood cell (WBC) count of >= 4000 cells/ml3, a platelet count of >= 100,000 cells/ml3, a serum bilirubin <= the institutional upper limit of normal, a serum serum glutamic-oxaloacetic transaminase (SGOT) or serum glutamic-pyruvic transaminase (SGPT) of <= 2.5 times the institutional upper limit of normal, and a serum creatinine of <= 2.0 times the institutional upper limit of normal.
* A post-prostatectomy pelvic computerized tomography (CT) scan, within 16 weeks prior to randomization, must reveal no evidence of metastatic disease.
* Patients must sign a study-specific informed consent form.
* Patients with prior invasive cancers are eligible if disease free for at least 5 years; prior or concurrent basal or squamous cell skin cancer is eligible.

Conditions for Patient Ineligibility:

* Pathologic stage T2 (without positive inked resection margin) or less except as stated in Section 3.1.1.1.
* Pathologic lymph node stage of pN1 or greater.
* An entry serum PSA of > 4.0ng/ml.
* Patients with persistant urinary extravasation after prostatectomy.
* Patients who have been previously treated with any hormonal therapy after prostatectomy.
* Patients who have previously been treated with radiation therapy or biologic therapy for prostate cancer.
* Karnofsky performance status < 80.
* Treatment start > 4 weeks after randomization.
* Prior chemotherapy for any reason.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 840 (Actual)
Dates: Start 1998-02; Primary Completion 2015-08 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William U. Shipley, MD, Principal Investigator — Massachusetts General Hospital and Harvard Medical School, Boston; Himanshu R Lukka, MD, Study Chair — Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, ON; Pierre P Major, MD, Study Chair — Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, ON; Niall M Heney, MD, Study Chair — Massachusetts General Hospital and Harvard Medical School, Boston; David J Grignon, MD, Study Chair — Indiana University, Indianapolis
Locations (240):
- United States (221):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Comprehensive Cancer Institute of Huntsville, Huntsville, Alabama
  - Huntsville Hospital System, Huntsville, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Alabama Oncology, LLC, Montgomery, Alabama
  - Radiation Oncology Associates of West Alabama, Tuscaloosa, Alabama
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Mount Diablo Medical Center, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Saint Agnes Cancer Center, Fresno, California
  - California Cancer Center, Fresno, California
  - Sutter Health West Cancer Research Group, Greenbrae, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Huntington Cancer Center, Pasadena, California
  - Cancer Care Center, Pomona, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - Radiation Medical Group, Inc., San Diego, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Saint Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Hospital of St. Raphael, New Haven, Connecticut
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - University of Florida Health Science Center, Gainesville, Florida
  - Florida Radiation Oncology Group, Jacksonville, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Sarasota Radiation and Medical Oncology Center, Sarasota, Florida
  - Tallahassee Memorial Healthcare, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical Center/John B. Amos Community Cancer Center, Columbus, Georgia
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - St. John's Medical Center, Anderson, Indiana
  - Bloomington Hospital, Bloomington, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Clarian Health Partners Inc., Indianapolis, Indiana
  - Regional Cancer Center, Indianapolis, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - Cancer Center at Lexington Clinic, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Louisville Radiation Oncology, Louisville, Kentucky
  - Merle M. Mahr Cancer Center, Madisonville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - Nebraska Health System, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Cooper Cancer Institute, Camden, New Jersey
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Atlantic City Medical Center, Pomona, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Capital Health System at Mercer, Trenton, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Associated Radiologists, P.A., Warren Township, New Jersey
  - Radiation Oncology Associates of Albuquerque, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Finger Lakes Radiation Oncology Center, Clifton Springs, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Riverhill Radiation Oncology, Yonkers, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Northeast Medical Center, Concord, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Barrett Cancer Center, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - St. Anthony Hospital, Oklahoma City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - St. John Health System, Tulsa, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Cancer Center, East Stroudsburg, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Wilkes Barre General Hospital, Wilkes-Barre, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Roger Williams Medical Center/BUSM, Providence, Rhode Island
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Bayshore Medical Center, Pasadena, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - RMH Regional Cancer Center, Harrisonburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Bon-Secours - St. Mary's Hospital, Richmond, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center, Wheeling, West Virginia
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - All Saints Cancer Center, Racine, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Canada (19):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Shipley WU, Seiferheld W, Lukka HR, Major PP, Heney NM, Grignon DJ, Sartor O, Patel MP, Bahary JP, Zietman AL, Pisansky TM, Zeitzer KL, Lawton CA, Feng FY, Lovett RD, Balogh AG, Souhami L, Rosenthal SA, Kerlin KJ, Dignam JJ, Pugh SL, Sandler HM; NRG Oncology RTOG. Radiation with or without Antiandrogen Therapy in Recurrent Prostate Cancer. N Engl J Med. 2017 Feb 2;376(5):417-428. doi: 10.1056/NEJMoa1607529. PMID 28146658
- [Derived] Brodowsky EC, Sood A, Butaney M, Majdalany SE, Stephens A, Corsi N, Piontkowski AJ, Rakic I, Jamil M, Dalela D, Peabody JO, Rogers CG, Abdollah F. Time to second biochemical recurrence as a prognostic indicator in postprostatectomy patients who undergo salvage radiation therapy: An RTOG 9601 based post hoc analysis. Prostate. 2023 Jan;83(1):64-70. doi: 10.1002/pros.24436. Epub 2022 Sep 19. PMID 36120850
- [Derived] Modonutti D, Majdalany SE, Corsi N, Li P, Sood A, Dalela D, Jamil ML, Hwang C, Menon M, Rogers CG, Trinh QD, Novara G, Abdollah F. A novel prognostic model predicting overall survival in patients with metastatic castration-resistant prostate cancer receiving standard chemotherapy: A multi-trial cohort analysis. Prostate. 2022 Sep;82(13):1293-1303. doi: 10.1002/pros.24403. Epub 2022 Jul 5. PMID 35790016
- [Derived] Jackson WC, Tang M, Schipper MJ, Sandler HM, Zumsteg ZS, Efstathiou JA, Shipley WU, Seiferheld W, Lukka HR, Bahary JP, Zietman AL, Pisansky TM, Zeitzer KL, Hall WA, Dess RT, Lovett RD, Balogh AG, Feng FY, Spratt DE. Biochemical Failure Is Not a Surrogate End Point for Overall Survival in Recurrent Prostate Cancer: Analysis of NRG Oncology/RTOG 9601. J Clin Oncol. 2022 Sep 20;40(27):3172-3179. doi: 10.1200/JCO.21.02741. Epub 2022 Jun 23. PMID 35737923
- [Derived] Feng FY, Huang HC, Spratt DE, Zhao SG, Sandler HM, Simko JP, Davicioni E, Nguyen PL, Pollack A, Efstathiou JA, Dicker AP, Todorovic T, Margrave J, Liu YS, Dabbas B, Thompson DJS, Das R, Dignam JJ, Sweeney C, Attard G, Bahary JP, Lukka HR, Hall WA, Pisansky TM, Shah AB, Pugh SL, Shipley WU, Tran PT. Validation of a 22-Gene Genomic Classifier in Patients With Recurrent Prostate Cancer: An Ancillary Study of the NRG/RTOG 9601 Randomized Clinical Trial. JAMA Oncol. 2021 Apr 1;7(4):544-552. doi: 10.1001/jamaoncol.2020.7671. PMID 33570548
- [Derived] Dess RT, Sun Y, Jackson WC, Jairath NK, Kishan AU, Wallington DG, Mahal BA, Stish BJ, Zumsteg ZS, Den RB, Hall WA, Gharzai LA, Jaworski EM, Reichert ZR, Morgan TM, Mehra R, Schaeffer EM, Sartor O, Nguyen PL, Lee WR, Rosenthal SA, Michalski JM, Schipper MJ, Dignam JJ, Pisansky TM, Zietman AL, Sandler HM, Efstathiou JA, Feng FY, Shipley WU, Spratt DE. Association of Presalvage Radiotherapy PSA Levels After Prostatectomy With Outcomes of Long-term Antiandrogen Therapy in Men With Prostate Cancer. JAMA Oncol. 2020 May 1;6(5):735-743. doi: 10.1001/jamaoncol.2020.0109. PMID 32215583
- Available data/document: Individual Participant Data Set: NCT00002874 — https://nctn-data-archive.nci.nih.gov/ — Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive.

RESULTS

PARTICIPANT FLOW:
Groups:
- Bicalutamide: Radiation therapy (64.8 Gy) + bicalutamide (150 mg daily 2 years)
- Placebo: Radiation therapy (64.8 Gy) + placebo (daily 2 years)
Period: Overall Study
Arm/Group | Bicalutamide | Placebo
Started | 421 | 419
Completed (Subjects with data available for the primary analysis are considered to have completed the study.) | 376 | 384
Not Completed | 45 | 35
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 44 | 34

BASELINE CHARACTERISTICS:
Population: Eligible patients who have not withdrawn
Groups:
- Total: Total of all reporting groups
Arm/Group | Bicalutamide | Placebo | Total
Number analyzed (Participants) | 376 | 384 | 760
Age, Continuous [Median (Full Range); unit: years] | 65 [45 to 81] | 65 [40 to 83] | 65 [40 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 376 | 384 | 760

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (12-year Rates Reported)
Description: Overall survival rates were estimated by the Kaplan-Meier method, with failure defined as death by any cause. Four-year follow-up was required of all patients, twelve-year rates are reported. Four-year follow-up was required of all patients, but twelve-year rates were reported.
  Patients are followed until death.
Time Frame: From date of randomization to 12 years.
Population: Eligible patients who did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Bicalutamide
Number analyzed (Participants) | 394 | 376
percentage of participants | 71.3 [66.5 to 76.0] | 76.3 [71.9 to 80.8]
Statistical Analysis 1: Comparison: Placebo vs Bicalutamide; Test type: Superiority; p = 0.020, Log Rank — One-sided significance level = 0.046 to preserve overall significance level of 0.05 for the study; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.59 to 0.98] — Stratifying variables were fixed covariates: prior hormone therapy (yes/no), entry prostate-specific antigen (PSA) (1.6-4.0 vs. 0.2-1.5), PSA nadir after surgery (< 0.5 vs. >= 0.5), positive surgical margins (yes/no). Reference level = placebo arm

2. Secondary Outcome: Non-Prostate Cancer Death (12-year Rates Reported)
Description: Non-prostate cancer death rates were estimated by the cumulative incidence method, with failure defined as any death that does not fall into the following categories: death due to prostate cancer or complications of protocol treatment (centrally reviewed), death with known progressive metastatic disease while on salvage hormone therapy, or death with a known rising PSA while on salvage hormone therapy. All other deaths are considered competing risks. Patients alive at time of analysis were censored. Any other death was treated as a competing risk. Four-year follow-up was required of all patients, but twelve-year rates were reported.
  Patients are followed until death. "Non-Prostate cancer death" is a more accurate wording for the protocol endpoint of "non-disease-specific survival", and matches the protocol definition.
Time Frame: From date of randomization to 12 years.
Population: Eligible patients who did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Bicalutamide
Number analyzed (Participants) | 376 | 384
percentage of participants | 15.3 [11.8 to 19.3] | 17.9 [14.0 to 22.1]
Statistical Analysis 1: Comparison: Placebo vs Bicalutamide; Test type: Superiority; p = 0.289, Gray's test; One-sided test; Cox Proportional Hazard = 1.10, 95% CI 2-sided [0.79 to 1.53]; Reference level = placebo arm

3. Secondary Outcome: Second PSA Recurrence (12-year Rates Reported)
Description: Second PSA recurrence (SPSAR) rates (i.e. first PSA failure on study) were estimated by the cumulative incidence method, with failure defined as the first occurrence of one of the following events: 1. Increase in PSA following protocol treatment according to the following criteria met during protocol treatment: If PSA dropped to undetectable level (<0.2 ng/ml) during protocol treatment (PT) then failure = increase after PT to >= 0.5 ng/ml ; If PSA decreased to a detectable level (≥ 0.2 ng/ml) during PT, then failure = increase PT of >= 0.3 ng/ml above the lowest detectable level; If PSA did not decrease during PT then failure = increase in PSA after PT of >= 0.5 ng/ml above entry PSA level. 2. The start of salvage hormone therapy. Patients alive without SPSAR at time of analysis were censored. Death without SPSAR was treated as a competing risk. Four-year follow-up was required of all patients, but twelve-year rates were reported. Patients are followed until death.
Time Frame: From date of randomization to 12 years.
Population: Eligible patients who did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Bicalutamide
Number analyzed (Participants) | 376 | 384
percentage of participants | 67.9 [62.7 to 72.5] | 44.0 [38.8 to 49.1]
Statistical Analysis 1: Comparison: Placebo vs Bicalutamide; Test type: Superiority; p < 0.001, Gray's test; One-sided test; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.40 to 0.58] — Reference level = placebo arm

4. Secondary Outcome: Third PSA Recurrence (12-year Rates Reported)
Description: Third PSA recurrence rates (i.e. second PSA failure on study) were estimated by the cumulative incidence method, with failure defined as PSA value of 0.5ng/ml or higher or any disease progression after starting salvage hormone therapy. Patients alive without third PSA recurrence at time of analysis were censored. Death without third PSA recurrence was treated as a competing risk. Four-year follow-up was required of all patients, but twelve-year rates were reported. Patients are followed until death.
Time Frame: From start of salvage hormone therapy to 12 years.
Population: Eligible patients who did not withdraw consent and who started salvage hormone therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Bicalutamide
Number analyzed (Participants) | 167 | 111
percentage of participants | 80.7 [73.2 to 86.3] | 84.2 [75.0 to 90.3]
Statistical Analysis 1: Comparison: Placebo vs Bicalutamide; Test type: Superiority; p = 0.213, Gray's test; One-sided test; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.85 to 1.46] — Reference level = placebo arm

5. Secondary Outcome: PSA Complete Response at End of Protocol Treatment
Description: Complete response is defined as a drop in PSA on protocol treatment to less than 0.2 ng/ml. Note that when the study opened many institutions could not detect PSA < 05 ng/ml.
Time Frame: End of protocol treatment, which is planned to last for two years
Population: Eligible patients who did not withdraw consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Bicalutamide
Number analyzed (Participants) | 376 | 384
Participants | 259 | 360
Statistical Analysis 1: Comparison: Placebo vs Bicalutamide; Test type: Superiority; p < 0.001, Chi-squared

6. Secondary Outcome: Distant Failure (12-year Rates Reported)
Description: Distant failure rates were estimated by the cumulative incidence method, with failure defined as the first occurrence of distant failure. Patients alive without distant metastases at time of analysis were censored. Death without distant metastasis was treated as a competing risk. Four-year follow-up was required of all patients, but twelve-year rates were reported. Patients are followed until death.
Time Frame: From date of randomization to 12 years.
Population: Eligible patients who did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Bicalutamide
Number analyzed (Participants) | 376 | 384
percentage of participants | 23.0 [18.8 to 27.5] | 14.5 [11.1 to 18.5]
Statistical Analysis 1: Comparison: Placebo vs Bicalutamide; Test type: Superiority; p = 0.002, Gray's test; One-sided test; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.46 to 0.87] — Reference level = placebo arm

7. Secondary Outcome: Prostate Cancer Death (12-year Rates Reported)
Description: Prostate cancer death rates were estimated by the cumulative incidence method, with failure defined as death due to prostate cancer or complications of protocol treatment (centrally reviewed), death with known progressive metastatic disease while on salvage hormone therapy, or death with a known rising PSA while on salvage hormone therapy. Patients alive at time of analysis were censored. Any other death was treated as a competing risk. Four-year follow-up was required of all patients, but twelve-year rates were reported. Patients are followed until death. "Prostate cancer death" is a more accurate wording for the protocol endpoint of "disease-specific survival", and matches the protocol definition.
Time Frame: From date of randomization to 12 years.
Population: Eligible patients who did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Bicalutamide
Number analyzed (Participants) | 376 | 384
percentage of participants | 13.4 [10.1 to 17.2] | 5.8 [3.6 to 8.6]
Statistical Analysis 1: Comparison: Placebo vs Bicalutamide; Test type: Superiority; p < 0.001, Gray's test; One-sided test; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.32 to 0.74] — Reference level = placebo arm

8. Secondary Outcome: Progression-free Survival (12-year Rates Reported)
Description: Progress-free survival rates were estimated by the Kaplan-Meier method, with failure defined as the first occurrence of PSA failure, local, regional or distant failure, or death from any cause. Patients alive without progression at time of analysis were censored. Four-year follow-up was required of all patients, but twelve-year rates were reported. Patients are followed until death. "Progression-free Survival" is more accurate wording for the protocol endpoint of "Freedom from Progression", and matches the protocol definition.
Time Frame: From date of randomization to 12 years.
Population: Eligible patients who did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Bicalutamide
Number analyzed (Participants) | 376 | 384
percentage of participants | 23.9 [19.4 to 28.4] | 38.8 [33.7 to 43.9]
Statistical Analysis 1: Comparison: Placebo vs Bicalutamide; Test type: Superiority; p < 0.001, Log Rank; One-side test; Cox Proportional Hazard = 0.60, 95% CI 2-sided [0.50 to 0.71]; Reference level = placebo arm

9. Secondary Outcome: Grade 3+ Toxicity
Description: Adverse events are graded using the Cooperative Group Common Toxicity Criteria and the Radiation Therapy Oncology Group (RTOG) Radiation Morbidity Scoring. Grade refers to severity, assigning Grades 1 through 5 based on this general guideline: Grade 0 None, Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related toxicity. Toxicities reported to have occurred within 90 days from the start of radiotherapy are reported as "Acute Radiotherapy", all later toxicities are reported as "Hormone therapy and late radiotherapy toxicity". The highest grade toxicity event per subject is counted within each of these time periods. Four-year follow-up was required of all patients; patients are followed until death.
Time Frame: From date of randomization to four years.
Population: Eligible patients who started protocol treatment and did not withdraw consent.
Measure: Number; unit: participants
Arm/Group | Placebo | Bicalutamide
Number analyzed (Participants) | 374 | 382
participants
  Acute radiotherapy toxicity | 17 | 8
  Hormone therapy and late radiotherapy toxicity | 73 | 100
Statistical Analysis 1: Comparison: Placebo vs Bicalutamide; Acute radiotherapy toxicity; Test type: Superiority; p = 0.060, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs Bicalutamide; Hormone therapy and late radiotherapy toxicity; Test type: Superiority; p = 0.029, Chi-squared

ADVERSE EVENTS:
Description: Subjects who started protocol treatment are included. Subjects experiencing more than one of a given toxicity are counted only once for that toxicity. Adverse events were graded with a combination of the Cooperative Group Common Toxicity Criteria and RTOG Acute and Late Radiation Morbidity Scoring. Grade refers to severity of toxicity assigning Grades 1-5: Grade 0 None, Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related toxicity.
Arm/Group | Placebo | Bicalutamide
Serious Adverse Events (participants affected / at risk) | 84/382 | 97/374
Other Adverse Events (participants affected / at risk) | 346/382 | 374/374
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=382) | Bicalutamide (N=374)
Acute RT Toxicity: Hematologic: NOS (Blood and lymphatic system disorders) | 3 | 2
Hematologic: NOS (Blood and lymphatic system disorders) | 5 | 5
Cardiac: NOS (Cardiac disorders) | 18 | 6
Acute RT Toxicity: Bowel: NOS (Gastrointestinal disorders) | 1 | 3
Bowel/GI: NOS (Gastrointestinal disorders) | 10 | 8
Nausea/vomiting: NOS (Gastrointestinal disorders) | 1 | 1
Acute RT Toxicity: Other: NOS (General disorders) | 0 | 1
Other: NOS (General disorders) | 16 | 16
Pain: NOS (General disorders) | 2 | 6
Liver: NOS (Hepatobiliary disorders) | 2 | 1
Neurologic: NOS (Nervous system disorders) | 8 | 5
Acute RT Toxicity: Bladder: NOS (Renal and urinary disorders) | 4 | 11
Bladder/GU: NOS (Renal and urinary disorders) | 28 | 30
Impotence: NOS (Reproductive system and breast disorders) | 28 | 16
Dyspnea: NOS (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Skin-general: NOS (Skin and subcutaneous tissue disorders) | 2 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=382) | Bicalutamide (N=374)
Acute RT Toxicity: Hematologic: NOS (Blood and lymphatic system disorders) | 34 | 28
Hematologic: NOS (Blood and lymphatic system disorders) | 58 | 36
Cardiac: NOS (Cardiac disorders) | 21 | 10
Acute RT Toxicity: Bowel: NOS (Gastrointestinal disorders) | 232 | 235
Bowel/GI: NOS (Gastrointestinal disorders) | 192 | 168
Nausea/vomiting: NOS (Gastrointestinal disorders) | 19 | 12
Acute RT Toxicity: Other: NOS (General disorders) | 68 | 50
Other: NOS (General disorders) | 129 | 100
Pain: NOS (General disorders) | 54 | 65
Acute RT Toxicity: Skin: NOS (Injury, poisoning and procedural complications) | 87 | 88
Skin-within XRT field: NOS (Injury, poisoning and procedural complications) | 46 | 34
Neurologic: NOS (Nervous system disorders) | 23 | 26
Acute RT Toxicity: Bladder: NOS (Renal and urinary disorders) | 188 | 165
Bladder/GU: NOS (Renal and urinary disorders) | 232 | 222
Gynecomastia: NOS (Reproductive system and breast disorders) | 266 | 42
Impotence: NOS (Reproductive system and breast disorders) | 46 | 37
Skin-general: NOS (Skin and subcutaneous tissue disorders) | 49 | 15
Hot flashes: NOS (Vascular disorders) | 83 | 67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.